CLINICAL TRIAL: NCT05953662
Title: Safety and Efficacy of Reduced-port Laparoscopic Surgery for Patients Of Colon and Upper Rectal Cancer --an Open Label, Multicenter, Prospective Phase Ⅱ Study
Brief Title: Safety and Efficacy of Reduced-port Laparoscopic Surgery for Patients Of Colon and Upper Rectal Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2023044
Record Dates: First submitted 2023-06-28; First posted 2023-07-20 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Neoplasm
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reduced-port laparoscopic surgery (Experimental): locations of trocars: A 10mm trocar is placed in the supraumbilical or subumbilicus as an observation port, and the surgeon inserts a 10mm trocar and a 5mm trocar on the ipsilateral side of the patient according to the intraoperative situation, as the main operation port and the secondary operation port, and the positions of the trocars follow the principle that the lesion is located at the triangular apex of the two trocars.
  Interventions: Procedure: Reduced-port laparoscopic surgery
- conventional laparoscopic surgery (Active Comparator): locations of trocars: A 10mm trocar is placed in the supraumbilicus or subumbilicus as an observation port, and the surgeon inserts a 10mm trocar and a 5mm trocar in a suitable position according to the intraoperative situation as the main operation port and the secondary operation port. The assistant places two 5mm trocars in the appropriate position as the assistant operation port.
  Interventions: Procedure: conventional laparoscopic surgery

INTERVENTIONS:
Procedure: Reduced-port laparoscopic surgery — compare different operational styles of colon and upper rectal cancer
  Arms: Reduced-port laparoscopic surgery
Procedure: conventional laparoscopic surgery — conventional laparoscopic surgery
  Arms: conventional laparoscopic surgery

SUMMARY:
Colorectal cancer is the third most common malignant tumor. Radical resection is the mainstay of treatments for non-metastatic colorectal cancer. In case of traditional laparoscopic surgery, inexperienced assistants are likely to cause side injuries and interfere surgeon due to limited operating space. Reduced-port laparoscopic surgery has only 3 ports for surgeon and observer, and the surgeon completes the surgery independently, which increases the difficulty of the operation. However, reduced-port laparoscopy has some potential advantages and applications. Reduced-port laparoscopic surgery avoids the prolongation of the operation time and parainjury caused by inexperienced assistant. Reduced-port laparoscopy reduces some surgical incisions, resulting in less pain and faster recovery. Reduced-port laparoscopy also reduces the consumables, human resources and medical expenses. This study aims to evaluate the curative effect and safety of reduced-port laparoscopic surgery versus conventional laparoscopic surgery for resectable colorectal cancer.

DETAILED DESCRIPTION:
Colorectal cancer is the third most common malignant tumor. In 2020, there were nearly 1.9 million new cases worldwide, accounting for about 10% of all new malignant tumors, and the related death exceeded 900,000. In recent years, the incidence of colorectal cancer in our country has been rising rapidly year by year, with more than 400,000 new cases each year, leading China to the largest number of colorectal cancer cases in the world. For resectable non-metastatic colorectal cancer, radical surgical resection is the mainstay of treatments. Compared with the open surgery, the laparoscopic colorectal cancer resection has smaller wounds, faster postoperative recovery, and shorter hospital stay. The 10-year results of the COLOR trial showed similar DFS, OS, and recurrence rates between open and laparoscopic surgery for colon cancer. In another trial (COST study), 872 patients with colon cancer were randomly assigned to open surgery or laparoscopic-assisted colectomy for curative colon cancer. After a median follow-up of 7 years, the 5-year recurrence rates and the 5-year OS rates were similar.

Traditional laparoscopic colorectal cancer resection can be carried out smoothly by close cooperation between the surgeon and the assistant. However, inexperienced assistants are likely to cause parainjuries due to the opposite field of the view and the narrow operating space. In recent years, single-port laparoscopy gradually goes into service. However, it is easy to cause instrument conflicts, straight-line viewing angles, and lack of traction. Therefore, single-port surgery is extremely unergonomic and difficult for the surgeon. Reduced-port laparoscopic surgery has been selectively used in some colon cancer anticipants. Reduced-port laparoscopic surgery reduces or completely eliminates the assistant's operating ports, and the surgeon mainly relies on himself/herself to complete the exposure of the operative field. However, reduced-port laparoscopy has some potential advantages and applications. Reduced-port laparoscopic surgery is completed by the left and right hands of the surgeon, which is easier to coordinate, avoiding the prolongation of the operation time or even concomitant injury caused by the poor cooperation of the inexperienced assistant and the surgeon. Reduced-port laparoscopy reduces some surgical incisions, and extreme minimally invasive may result in less pain and faster recovery. From an economic point of view, the reduced-port laparoscopy reduces some surgical consumables and human resouce, leading to reduced cost of surgery.

In order to further explore the application of reduced-port laparoscopic surgery in patients with resectable colorectal cancer, the center plans to carry out a clinical study of 'reduced-port laparoscopic surgery versus traditional laparoscopic surgery for resectable colorectal cancer', aiming to evaluate the complications associated with perioperative surgery, R0 resection rate, 3-year disease-free survival rate, and 3-year overall survival rate.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years old;
2. Pathological diagnosis of colorectal adenocarcinoma (including high, medium and low-differentiated adenocarcinoma, excluded: mucinous adenocarcinoma, signet ring cell carcinoma);
3. Eastern Cooperative Oncology Group (ECOG) is 0-1 points;
4. Chest, whole abdomen, pelvic enhanced CT confirm colon or upper rectal cancer, without distant metastasis;
5. No other multiple primary tumors;
6. No organ dysfunction;
7. The patient and his/her family are able to understand the study protocol and are willing to participate in the study and sign informed consent.

Exclusion Criteria:

1. Age < 18, or > 80 years old;
2. Combined with simultaneous or heterogeneous (within 5 years) malignant tumors;
3. Patients with intestinal obstruction, intestinal perforation, intestinal bleeding, etc. who require emergency surgery;
4. Joint organ resection is required;
5. ASA Class IV or V;
6. Suffering from a serious mental illness;
7. Patients with severe emphysema, interstitial pneumonia or ischemic heart disease, etc. who cannot tolerate surgery;
8. Continuous systemic steroid therapy within 1 months;
9. Patients or families are unable to understand the conditions and objectives of this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
DFS rate | 1 year
  Disease-free survival rate

SECONDARY OUTCOMES:
Total opertaion time | through opertation completion, an average of 2 hours
  Time from surgery started to surgery ended
Intraoperative blood loss | through study completion, an average of 50 ml
  Blood loss during operation
Postoperative hospital stay | through anticipants discharged, an average of 7 days
  Day from operation finished to patient discharged
Postoperative complication rate | 30 days
  Any complication associated with operation based on Clavien-Dindo classification
Postoperative mortality | 30 days
  Death associated with operation
3 years DFS Rate | 3 years
  Disease-free survival rate
3 years OS Rate | 3 years
  Overall survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Jun Huang, MD, Principal Investigator — six affiliated hospital of Sun Yat-sen University
Locations (1):
- The Sixth Affiliated Hospital, Sun Yatsen University, Guangzhou, Guangdong, China